CLINICAL TRIAL: NCT02683291
Title: Sirolimus Associated With Tacrolimus at Low Doses in Elderly Kidney Transplant Patients: A Prospective Randomized Controlled Trial
Brief Title: Sirolimus Associated With Tacrolimus at Low Doses in Elderly Kidney Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Associação Médico Espírita de Botucatu (Other)
Responsible Party: Principal Investigator, Luis Gustavo Modelli de Andrade, Clinical Professor PhD, Associação Médico Espírita de Botucatu
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16966913.6.0000.5411
Record Dates: First submitted 2016-02-05; First posted 2016-02-17 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Disorder Related to Renal Transplantation; Cytomegalovirus Infections
Keywords: Kidney transplantation; sirolimus; cytomegalovirus; aged
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Sirolimus; Tacrolimus; Mycophenolic Acid; Prednisone; Basiliximab; thymoglobulin; Antilymphocyte Serum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tacrolimus + Mycophenolate (Active Comparator): The investigators wil be used tacrolimus (starting with 0.1 mg/kg twice daily adjusted to target serum levels by 4-8ng/ml at the third month and then 3-7ng/ml from the third month to the 12th month) and mycophenolate sodium 720 mg twice daily. A dose reduction of mycophenolate sodium to 720 mg/day will be accepted due to possible side effects of the drug.
  Prednisone 30 mg/day in the first month. Induction therapy consisted of basiliximab or thymoglobulin if panel reactivity class I greater than 50 %
  Interventions: Drug: tacrolimus; Drug: mycophenolate; Drug: Prednisone; Drug: Basiliximab; Drug: Thymoglobulin
- Tacrolimus + Sirolimus (Experimental): The investigators will be used tacrolimus (starting with 0.1 mg/kg twice daily adjusted to target serum levels by 4-8 ng/ml at the third month and then 3-7 ng/ml from the third month to the 12th month) and sirolimus 2 mg/day (adjusted serum levels at 4-8 ng/ml throughout the study period).
  Prednisone 30 mg/day in the first month. Induction therapy consisted of basiliximab or thymoglobulin if panel reactivity class I greater than 50 %
  Interventions: Drug: sirolimus; Drug: tacrolimus; Drug: Prednisone; Drug: Basiliximab; Drug: Thymoglobulin

INTERVENTIONS:
Drug: sirolimus
  Other Names: Rapamycin; Rapamune
  Arms: Tacrolimus + Sirolimus
Drug: tacrolimus
  Other Names: Prograf; FK506
Drug: mycophenolate
  Other Names: Myfortic; Mycophenolate Sodium
  Arms: Tacrolimus + Mycophenolate
Drug: Prednisone — Prednisone 30mg/day
  Other Names: Meticorten
Drug: Basiliximab — Basiliximab 20mg (first and fourth day) if panel reactivity class I less than 50 %
  Other Names: Simulect
Drug: Thymoglobulin — Thymoglobulin at a dose of 1mg/kg for 5 days if panel reactivity class I greater than 50 %
  Other Names: antithymocyte globulin

SUMMARY:
There is no consensus on the best immunosuppressive regimen in elderly people. The aim of this study will be to evaluate the efficacy of sirolimus associated with tacrolimus in elderly kidney transplant recipients. The investigators will conduct a single-center prospective randomized study comparing the combination of tacrolimus with sirolimus at reduced dose rate (tacrolimus + sirolimus group) against tacrolimus with mycophenolate (tacrolimus + mycophenolate group). The investigators will include all kidney transplant patients over 60 years of age. The investigators will evaluate estimated glomerular filtration rate and incidence of cytomegalovirus in 12 month follow-up.

DETAILED DESCRIPTION:
Study Design

This will be a single-center, prospective, 12-month randomized controlled trial aiming to compare sirolimus associated with tacrolimus in elderly renal transplant patients as to safety and incidence of cytomegalovirus (CMV) infection.

Treatments

In the control group (Tacrolimus + Mycophenolate) the investigators will use tacrolimus (starting with 0.1 mg/kg twice daily adjusted to target serum levels by 4-8ng/ml at the third month and then 3-7ng/ml from the third month to the 12th month) and mycophenolate sodium 720 mg twice daily. A dose reduction of mycophenolate sodium to 720 mg/day will be accepted due to possible side effects of the drug.

In the treatment group (Tacrolimus + sirolimus) the investigators will use tacrolimus (starting with 0.1 mg/kg twice daily adjusted to target serum levels by 4-8 ng/ml at the third month and then 3-7 ng/ml from the third month to the 12th month) and sirolimus 2 mg/day (adjusted serum levels at 4-8 ng/ml throughout the study period).

In all groups, patients will receive prednisone 30 mg/day (in the first month with weekly reductions up to 5 mg/day at the end of the second month). Induction therapy consisted of basiliximab or antithymocyte globulin (Thymoglobulin, Genzyme®). Thymoglobulin will be used in patients with panel reactivity class I greater than 50 % (at a dose of 1mg/kg for 5 days).

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged more than 60 years and recipients of compatible renal transplant

Exclusion Criteria:

1. Receptors of multiple organs;
2. non-heart beating donors;
3. donors aged under 5 or over 65 years;
4. Patients with body mass index greater than 35

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in estimated glomerular filtration rate from baseline | Baseline, 1 month, 3 months, 6 months and 12 months
  The primary end-point will be evaluated the estimated glomerular filtration rate (eGFR) over 12 months of renal transplantation. The investigators will be measure the change in eGFR during 12 month follow-up. Glomerular filtration rate will be estimated by the MDRD equation (Modification of Diet in Renal Disease).

SECONDARY OUTCOMES:
Incidence of cytomegalovirus Infection (CMV) | Weekly from baseline until the third month. After in 4, 5, 6, 8, 10 and 12 months.
  The secondary end-point will be evaluated the incidence of cytomegalovirus (CMV) infection. CMV infection will be defined based on detection of CMV viral replication (CMV pp65 antigenemia more than zero) in asymptomatic patients. CMV disease will be defined based on the evidence of CMV infection with related symptoms. For the positive cases treatment will be carried out with ganciclovir 5 mg/kg/day twice daily adjusted for renal function for a minimum of 14 days.

IPD SHARING:
Plan to Share IPD: No